CLINICAL TRIAL: NCT02411396
Title: Patient Centered Outcomes Research Institute (PCORI) ESCAPED Study: Comparison of Patient Centered Outcomes for People With SCD in the Acute Care Setting
Brief Title: Comparison of Patient Centered Outcomes for People With Sickle Cell Disease in the Acute Care Setting
Acronym: ESCAPED
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00054029; PCORI-1403-11888 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2015-03-30; First posted 2015-04-08 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients With SCD: Patients treated for uncomplicated VOC in ICs and EDs.

SUMMARY:
The Emergency Department has been the standard location where patients with Sickle Cell Disease (SCD) go to seek care for the treatment of acute painful events. Vaso- Occlusive Crisis (VOC) is the most common complication of SCD,

The purpose of this study is to compare patient centered outcomes for patients being treated for an uncomplicated VOC in Infusion Centers (IC) and Emergency Departments (ED) in four locations around the United States.

DETAILED DESCRIPTION:
Emergency Department care is marked by long delays, lack of efficacy, and conflict. A sub-specialty Infusion Center staffed by expert clinicians and delivering individualized care can improve care quality while reducing costs. The study will examine whether care provided in an Infusion Center (IC) is more patient centered and efficient than care provided in an Emergency Department (ED) for adults with Sickle Cell Disease (SCD) and uncomplicated Vaso-Occlusive Crisis (VOC).

Sites will prospectively enroll patients in VOC seen in participating centers from either the EDs or the ICs. Specific data from the acute visits (e.g. Times of arrival, time to first dose of analgesic, etc) will be captured. This study will compare: pain management, disposition of subjects (home or admission) and patient experiences of care delivery in both settings. Subjects will complete surveys/questionnaires to asses subjects' experiences in the setting where care was provided.

The four sites to participate in the study are Baltimore, Maryland (Johns Hopkins Hospital), Cleveland, Ohio (Cleveland Medical Center), Milwaukee, Wisconsin (Medical College of Wisconsin), and Baton Rouge, Louisiana (Our Lady of the Lake Hospital). A maximum of 500 subjects will participate in the study. Participants will be enrolled for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Sickle Cell Disease patients who live within 60 miles of the study center or who already receive regular care at the participating centers.

Exclusion Criteria:

* Stable patients who have been on chronic transfusion therapy and have not had a painful episode within two years of enrollment.
* Patients who are pregnant.
* Patients who are unwilling or unable to sign consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with SCD inclusive of genotypes homozygous and compound heterozygous sickle hemoglobin. In the United States, SCD primarily afflicts African-American and Hispanic-American populations. Patients will be enrolled prior to a vaso-occlusive crisis and data will be collected from patients' acute visit(s) at either the Emergency Department or at an Infusion center (4 participating sites).
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lanzkron, MD, MHS, Principal Investigator — Johns Hopkins University, Division of Hematology
Locations (3):
- United States (3):
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Cleveland Medical Center at University Hospitals, Cleveland, Ohio
  - Medical College of Wisconsin, Blood Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hassell KL. Population estimates of sickle cell disease in the U.S. Am J Prev Med. 2010 Apr;38(4 Suppl):S512-21. doi: 10.1016/j.amepre.2009.12.022. PMID 20331952
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] McClish DK, Penberthy LT, Bovbjerg VE, Roberts JD, Aisiku IP, Levenson JL, Roseff SD, Smith WR. Health related quality of life in sickle cell patients: the PiSCES project. Health Qual Life Outcomes. 2005 Aug 29;3:50. doi: 10.1186/1477-7525-3-50. PMID 16129027
- [Background] Bediako SM. Predictors of employment status among African Americans with sickle cell disease. J Health Care Poor Underserved. 2010 Nov;21(4):1124-37. doi: 10.1353/hpu.2010.0945. PMID 21099066
- [Background] Lanzkron S, Carroll CP, Hill P, David M, Paul N, Haywood C Jr. Impact of a dedicated infusion clinic for acute management of adults with sickle cell pain crisis. Am J Hematol. 2015 May;90(5):376-80. doi: 10.1002/ajh.23961. Epub 2015 Feb 25. PMID 25639822
- [Background] Haywood C Jr, Tanabe P, Naik R, Beach MC, Lanzkron S. The impact of race and disease on sickle cell patient wait times in the emergency department. Am J Emerg Med. 2013 Apr;31(4):651-6. doi: 10.1016/j.ajem.2012.11.005. Epub 2013 Feb 4. PMID 23380119
- [Background] Lanzkron S, Carroll CP, Haywood C Jr. The burden of emergency department use for sickle-cell disease: an analysis of the national emergency department sample database. Am J Hematol. 2010 Oct;85(10):797-9. doi: 10.1002/ajh.21807. PMID 20730795
- [Derived] Lanzkron S, Little J, Wang H, Field JJ, Shows JR, Haywood C Jr, Saheed M, Proudford M, Robertson D, Kincaid A, Burgess L, Green C, Seufert R, Brooks J, Piehet A, Griffin B, Arnold N, Frymark S, Wallace M, Abu Al Hamayel N, Huang CY, Segal JB, Varadhan R. Treatment of Acute Pain in Adults With Sickle Cell Disease in an Infusion Center Versus the Emergency Department : A Multicenter Prospective Cohort Study. Ann Intern Med. 2021 Sep;174(9):1207-1213. doi: 10.7326/M20-7171. Epub 2021 Jul 6. PMID 34224261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There are a total of 483 adult patients with sickle cell disease (SCD) enrolled from the end of April 2015 to December, 2016. 145 from Johns Hopkins (JH), 101 from Case Western (CW), 110 from Our Lady of the Lake Hospital (OLL) and 127 from Blood Center of Wisconsin (BCW). Four hundred forty two patients have completed 18 months follow up
Groups:
- Vaso-Occlusive Crisis (VOC) in Patients With SCD: Patients treated for uncomplicated Vaso-Occlusive Crisis (VOC) in ICs and EDs.
Period: Overall Study
Arm/Group | Vaso-Occlusive Crisis (VOC) in Patients With SCD
Started (First participant enrolled on 4/30/2015 at Johns Hopkins) | 483
Completed | 442
Not Completed | 41
Not completed — Lost to Follow-up | 31
Not completed — Death | 10

BASELINE CHARACTERISTICS:
Groups:
- VOC in Patients With SCD: Patients treated for uncomplicated VOC in ICs and EDs.
Arm/Group | VOC in Patients With SCD
Number analyzed (Participants) | 483
Age, Categorical [Count of Participants; unit: Participants] — age of participant in years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 476
    >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 293
  Male | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 477
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 471
  White | 0
  More than one race | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 483

OUTCOME MEASURES:

1. Primary Outcome: Time (Minutes) From Arrival to Center to Time First Dose of Parenteral Pain Medication Administered
Description: Time is recorded from the time the patient arrives for pain treatment at either the ED or IC until the time the patient is dosed with pain medication administered parenterally. Guideline recommendations are that patients receive non-oral pain medication within 60 minutes of arrival.
Time Frame: Within 6 hours after arrival
Population: Not all participants enrolled in the study visited the ED or the IC for uncomplicated vaso-occlusive crisis. The total number of subjects analyzed exceeds the total number of subjects because the same subject could visit the ED or IC one or more times.
Measure: Mean (95% Confidence Interval); unit: minutes
Units Other Than Participants: number of visits
Groups:
- VOC in Patients With SCD Who Went to EDs: Patients treated for uncomplicated VOC in EDs.
- VOC in Patients With SCD Who Went to ICs: Patients treated for uncomplicated VOC in ICs
Arm/Group | VOC in Patients With SCD Who Went to EDs | VOC in Patients With SCD Who Went to ICs
Number analyzed (Participants) | 317 | 265
Number analyzed (number of visits) | 1558 | 1469
minutes | 125.3 [118.3 to 131.8] | 61.8 [59.3 to 64.3]
Statistical Analysis 1: Comparison: VOC in Patients With SCD Who Went to EDs vs VOC in Patients With SCD Who Went to ICs; This analysis is to compare outcome measure between ED or IC visits by using time varying propensity score method developed by our group to adjust imbalance of covariates between the two arms. Each patient can have multiple visits to the facility of choice; Test type: Other — In order to eliminate bias from the naïve estimation on the treatment effects due to the confounders, time varying propensity score model was developed. This balanced the covariates between the two arms at each single acute visit of each patient. A sub classification on the propensity scores was used to estimate the potential outcome for each arm and the average treatment effects (ATE). Bootstrapping was employed to estimate the standard error of ATE; Mean Difference (Final Values) = 124.6, 95% CI 2-sided [118.3 to 130.9], Standard Error of Mean 3.2

2. Secondary Outcome: Disposition From Acute Care Visit
Description: Odds for admission to the hospital versus discharge to home (ED vs IC)
Time Frame: Day 1 of admission
Population: as for outcome 1
Measure: Number; unit: number of visits
Units Other Than Participants: number of visits
Arm/Group | VOC in Patients With SCD Who Went to EDs | VOC in Patients With SCD Who Went to ICs
Number analyzed (Participants) | 317 | 265
Number analyzed (number of visits) | 1556 | 1468
number of visits
  Number of visits being hospitalized | 517 | 128
  Number of visits being sent home | 1039 | 1340
Statistical Analysis 1: Comparison: VOC in Patients With SCD Who Went to EDs vs VOC in Patients With SCD Who Went to ICs; Test type: Other — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.14, 95% CI 2-sided [4.13 to 6.41] — VOC in patients with SCD whom went to EDs represents the numerator, VOC in patients with SCD whom went to ICs represents the denominator for Odds Ratio

3. Secondary Outcome: Pain Reassessment Within 30 Minutes of First Dose of Parenteral Pain Medication Administered
Description: Odds of being re-assessed for pain within 30 minutes of receiving first dose of pain medication in ED vs IC. NHLBI guidelines recommend that patients are re-assessed for adequacy of pain management 30 minutes after receiving pain medication.
Time Frame: 30 minutes after administration
Population: as for outcome 1
Measure: Number; unit: number of visits
Units Other Than Participants: number of visits
Arm/Group | VOC in Patients With SCD Who Went to EDs | VOC in Patients With SCD Who Went to ICs
Number analyzed (Participants) | 317 | 265
Number analyzed (number of visits) | 1394 | 1455
number of visits
  Number of visits being reassessed in 30 mins | 287 | 544
  Number of visits not being reassessed in 30 mins | 1107 | 911
Statistical Analysis 1: Comparison: VOC in Patients With SCD Who Went to EDs vs VOC in Patients With SCD Who Went to ICs; Test type: Other — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.84 to 2.72] — VOC in patients with SCD whom went to ICs represents the numerator, VOC in patients with SCD whom went to EDs represents the denominator for Odds Ratio

4. Secondary Outcome: Patient Reported Satisfaction With Care Received
Description: Survey to capture patient satisfaction with the quality of care in either the ED or IC. Validated a new tool to assess satisfaction with care in the acute care setting. The new tool was developed based on existing tools that assessed several domains: adequacy of pain management, communication with providers, interpersonal aspects of care, provider competence, involvement of family/friends, and access to care. The final 15 item validated Patient Satisfaction with Pain Management in Sickle Cell Disease (SCD) (PSPS) scale was used to compare satisfaction of care comparing ED to IC acute visits. Overall mean satisfaction scores ranged from 0-7 with higher scores signifying greater satisfaction
Time Frame: within 72 hours of acute visit
Population: 207 participants completed the satisfaction survey after their first visit during the study time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- VOC in Patients With SCD Who Went to the ED: VOC in Patients with SCD that went to the ED
- VOC in Patients With SCD Who Went to the IC: VOC in patients with SCD that went to the IC
Arm/Group | VOC in Patients With SCD Who Went to the ED | VOC in Patients With SCD Who Went to the IC
Number analyzed (Participants) | 85 | 122
score on a scale | 4.8 (1.1) | 5.8 (1.0)

5. Secondary Outcome: Patient Reported Perception of Risk From Visit
Description: One question on the survey asked patients to rate the overall level of medical safety they felt during their visit to the ED or IC. Choices for responses: Excellent, Very Good, Good, Fair or Poor. Excellent and Very Good were determined as having greater feelings of overall safety while patients who chose Good, Fair or Poor were determined having lesser feelings of overall safety.
Time Frame: within 72 hours of acute visit
Population: Only 205 patients completed the perception of risk question at the first visit to either the ED or the IC.
Measure: Count of Participants; unit: Participants
Groups:
- VOC in Patients With SCD Who Went to ED: Patients treated for uncomplicated VOC in EDs
- VOC in Patients With SCD Who Went to IC: Patients treated for uncomplicated VOC in ICs
Arm/Group | VOC in Patients With SCD Who Went to ED | VOC in Patients With SCD Who Went to IC
Number analyzed (Participants) | 87 | 118
Participants
  Greater feelings of overall medical safety | 43 | 98
  Lesser feelings of overall safety | 44 | 20

ADVERSE EVENTS:
Time Frame: Participants were followed for 18 months
Description: No adverse events were collected since observational study.
Arm/Group | VOC in Patients With SCD
All-Cause Mortality (participants affected / at risk) | 10/483
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02411396/Prot_SAP_000.pdf